CLINICAL TRIAL: NCT00049400
Title: A Phase I Pharmacokinetic Study Of Epothilone B Analogue BMS-247550 (NSC 710428D) In Patients With Advanced Malignancies And Varying Levels Of Liver Dysfunction
Brief Title: S0355 Ixabepilone in Treating Patients With Advanced Solid Tumors or Lymphomas and Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0355; U01CA076642 (NIH); P30CA016087 (NIH); S0355 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; intraocular lymphoma; primary central nervous system lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1, 2, or 3 follicular lymphoma; recurrent mantle cell lymphoma; small intestine lymphoma; stage IV adult diffuse large cell or mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma or Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1, 2, or 3 follicular lymphoma; stage IV mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of MALT; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult Burkitt lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): Single-arm, dose-escalation of BMS-247550
  Interventions: Drug: BMS-247550

INTERVENTIONS:
Drug: BMS-247550 — BMS-247550 as a 3-hour infusion on Day 1 of a three-week cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of ixabepilone in treating patients with advanced solid tumors or lymphomas and liver dysfunction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the levels of hepatic impairment at which dose modifications of ixabepilone are required in patients with advanced solid tumors or lymphomas and varying levels of liver dysfunction.
* Determine the effect of hepatic dysfunction on the plasma pharmacokinetics of this drug in these patients.
* Determine the toxic effects of this drug at varying levels of hepatic dysfunction in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to liver function (normal vs mild dysfunction vs moderate dysfunction vs severe dysfunction).

Patients receive ixabepilone IV over 3 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 6 but no more than 12 patients are treated at the recommended phase II dose.

Patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 12-84 patients (6-12 for stratum 1; 2-18 for stratum 2; 2-24 for stratum 3; and 2-30 for stratum 4) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor or lymphoma for which standard curative or palliative measures do not exist or are no longer effective

  * Pathological confirmation of diagnosis not required in patients with liver mass, raised alpha-fetoprotein levels (at least 500 ng/mL), and positive serology for hepatitis consistent with a diagnosis of hepatocellular carcinoma
  * Any solid tumor or lymphoma tumor type eligible
  * Must have had thoracic and upper abdominal CT scan, including entire liver and adrenals, within 28 days before study entry
* Patients with glioma or brain metastases must be on a stable dose of corticosteroids and be seizure-free for the past month

  * Prior whole brain or gamma knife radiotherapy required for known brain metastases
  * No unstable or untreated (non-irradiated) brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No active hemolysis

Hepatic

* See Disease Characteristics
* Patients with biliary obstruction for which a shunt has been placed are allowed if shunt is in place for at least 10 days and liver function is stable
* Abnormal liver function (bilirubin and SGOT) allowed regardless of cause (metastases or other causes)
* No evidence of biliary sepsis

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* No concurrent uncontrolled illness
* No ongoing or active infection
* No uncontrolled diarrhea
* No peripheral neuropathy grade II or greater
* No psychiatric illness or social situation that would preclude study compliance
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy for malignancy

Chemotherapy

* More than 2 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy for malignancy

Endocrine therapy

* See Disease Characteristics
* No concurrent oral contraceptives
* No concurrent hormone therapy for malignancy

  * Concurrent luteinizing hormone-releasing hormone agonists allowed

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy for malignancy

Surgery

* More than 2 weeks since prior major surgery

Other

* Recovered from prior therapy
* No concurrent medications that are known to be inhibitors of CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2003-10; Primary Completion 2006-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
dose defining | Treatment delays >2 weeks constitute a DLT

SECONDARY OUTCOMES:
Progression | 30 days after going off study
  20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline.
Symptomatic deterioration | 30 days after going off study
  Global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Davies, MD, Principal Investigator — University of California, Davis; Chris H. Takimoto, MD, PhD, Principal Investigator — Institute for Drug Development
Locations (23):
- United States (23):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington

REFERENCES:
- [Result] Takimoto CH, Liu PY, Lenz H, et al.: A phase I pharmacokinetic (PK) study of the epothilone B analogue, ixabepilone (BMS-247550) in patients (pts) with advanced malignancies and varying degrees of hepatic impairment. A SWOG Early Therapeutics Committee and NCI Organ Dysfunction Working Group Trial. [Abstract] J Clin Oncol 24 (Suppl 18): A-2004, 2006.